CLINICAL TRIAL: NCT00428194
Title: Erlotinib in Combination With Cisplatin as Radiosensitizing Agents in Women Receiving Radiation Therapy for Locally Advanced Squamous Cell Carcinoma of the Cervix; A Phase I Trial
Brief Title: Erlotinib, Cisplatin, and Radiation Therapy in Treating Patients With Stage IB-Stage IVA Cervical Cancer
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Withdrawn due to lack of accrual
Sponsor: Masonic Cancer Center, University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2006LS019; UMN-0604M84827 (Other: IRB, University of Minnesota)
Record Dates: First submitted 2007-01-25; First posted 2007-01-29 (Estimated); Last update posted 2017-11-29 (Actual); Status verified 2017-11

CONDITIONS: Cervical Cancer
Keywords: stage IIA cervical cancer; stage IB cervical cancer; stage IIB cervical cancer; stage III cervical cancer; stage IVA cervical cancer; cervical squamous cell carcinoma
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Cisplatin; Erlotinib Hydrochloride; Radiotherapy; Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Cohort 1 (Experimental): Erlotinib 100 mg/day by mouth beginning on day 1 of radiotherapy (RT) and cisplatin dosing (40 mg/m^2 intravenous every 7 days during RT) and continuing daily through radiation
  Interventions: Drug: cisplatin; Drug: erlotinib hydrochloride; Procedure: radiation therapy
- Cohort 2 (Experimental): Erlotinib 125 mg/day by mouth beginning on day 1 of radiotherapy (RT) and cisplatin dosing (40 mg/m^2 intravenous every 7 days during RT) and continuing daily through radiation
  Interventions: Drug: cisplatin; Drug: erlotinib hydrochloride; Procedure: radiation therapy
- Cohort 3 (Active Comparator): Erlotinib 150 mg/day by mouth beginning on day 1 of radiotherapy (RT) and cisplatin dosing (40 mg/m^2 intravenous every 7 days during RT) and continuing daily through radiation
  Interventions: Drug: cisplatin; Drug: erlotinib hydrochloride; Procedure: radiation therapy

INTERVENTIONS:
Drug: cisplatin — 40 mg/m^2 every 7 days during radiation
  Other Names: cisplatinum; CDDP
Drug: erlotinib hydrochloride — Erlotinib escalating dose per schedule - 100, 125 and 150 mg/m^2 by mouth once a day beginning day 1.
  Other Names: Tarceva(R)
Procedure: radiation therapy — standard (fixed) doses of pelvic irradiation (as determined by their radiation oncologist)
  Other Names: irradiation

SUMMARY:
RATIONALE: Erlotinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Drugs used in chemotherapy, such as cisplatin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Radiation therapy uses high-energy x-rays to kill tumor cells. Erlotinib and cisplatin may make tumor cells more sensitive to radiation therapy. Giving erlotinib together with cisplatin and radiation therapy may kill more tumor cells.

PURPOSE: This phase I trial is studying the side effects and best dose of erlotinib when given together with cisplatin and radiation therapy in treating patients with stage IB, stage II, stage III, or stage IVA cervical cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the maximum tolerated dose of erlotinib hydrochloride when administered with cisplatin and pelvic radiotherapy in patients with stage IB-IVA squamous cell carcinoma of the cervix.

Secondary

* Determine the toxicity profile of this regimen.

OUTLINE: This is a multicenter, open-label, dose-escalation study of erlotinib hydrochloride.

Patients receive oral erlotinib hydrochloride once daily on days 1-35 and cisplatin IV on days 1, 8, 15, 22, and 29. Patients also undergo radiotherapy daily, 5 days a week, for approximately 5 weeks concurrently with chemotherapy.

Cohorts of 3-6 patients receive escalating doses of erlotinib hydrochloride until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose proceeding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity.

After completion of study treatment, patients are followed at 6 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of squamous cell carcinoma of the cervix

  * Stage IB-IVA disease
* Scheduled to undergo standard radiotherapy and receive weekly cisplatin
* ECOG performance status 0-2
* Not pregnant
* Negative pregnancy test
* Fertile patients must use effective contraception during and for ≥ 1 week after completion of study treatment
* Must be able to take oral medication

Exclusion Criteria:

* Malabsorption syndrome
* Serious underlying medical condition that would impair the ability of patient to receive treatment
* Known hypersensitivity to erlotinib hydrochloride
* Psychological, familial, sociological, or geographical conditions that would preclude study compliance
* Less than 21 days since prior nonapproved or investigational drugs
* Prior chemotherapy
* Prior radiotherapy
* Prior anti-epidermal growth factor receptor treatment
* Prior gastrointestinal surgery that limits absorption (i.e., requiring total parenteral nutrition)
* Concurrent use of any of the following agents and therapies:

  * Other antineoplastic or antitumor agents
  * Other chemotherapy
  * Other investigational agents
  * Radiotherapy
  * Immunotherapy
  * Anticancer hormonal therapy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2007-01; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose of erlotinib hydrochloride | Day 14

SECONDARY OUTCOMES:
Toxicity | 4-6 Weeks Post Last Study Dose

CONTACTS AND LOCATIONS:
Overall Officials: Levi S. Downs, MD, Study Chair — Masonic Cancer Center, University of Minnesota
Locations (1):
- University of Minnesota Cancer Center, Minneapolis, Minnesota, United States